CLINICAL TRIAL: NCT00283127
Title: Home Sampling Versus Conventional Sampling for Screening of Urogenital Chlamydia Trachomatis in Young Men and Women. - A Randomised Control Trial
Brief Title: Home Sampling Versus Conventional Sampling for Screening of Urogenital Chlamydia Trachomatis in Young Men and Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2.2005.1223
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2009-01

CONDITIONS: Chlamydia Trachomatis; Mass Screening
Keywords: Chlamydia trachomatis; Mass screening; Home sampling; Urine test
MeSH Terms: interventions — Urinalysis

INTERVENTIONS:
Procedure: Home sampling (urine test) for uro-genital C.trachomatis.

SUMMARY:
Urogenital Chlamydia trachomatis infection is the most common bacterial sexually transmitted infection in Norway. Urogential C.trachomatis infection can easily be treated with antibiotics. However, left untreated it is a major cause of pelvic inflammatory disease (PID) that can lead to complications such as infertility, ectopic pregnancy and chronic pelvic pain in women. Most infections are asymptomatic and many do not seek the doctor for testing. Therefore cases remain undetected and untreated.We want to determine the efficacy and feasibility of screening for urogenital C. trachomatis infection with home sampling (intervention) compared to the current strategy of conventional sampling at the doctor's office (control) in identifying men and women aged 18-25 years with urogenital C.trachomatis infection (Part A). We also want to identify factors influencing the acceptability of home sampling for C.trachomatis infections (Part B)and determine factors associated with C.trachomatis infections (Part C).

DETAILED DESCRIPTION:
Study design The different objectives will be addressed through a complex design with several sub-studies.

Part A is a randomised control trial where we compare the intervention group who will be offered home-sampling and recieve a package by mail (containing information on urogenital C.trachomatis infections, sampling eqiupment for urine tests and a questionnaire) with a control group who will continue with todays system of conventional sampling at the doctores office (no intervention). The study population are all men and women between 18-25 years of age in Rogaland County in Norway. The population register will be used to randomly assigne to either the intervention group or the control group.The intervention group will be asked to take a urine sample and send this by mail to the laboratory for analysis within three months after the invitation, and to fill out and return a questionnaire. For the ones in the control group all samples(urethral or cervical swabs or urine samples)taken within the same three months will be sendt to the same laboratory. In this part of the study we will measure the yield ratio for the tested, diagnosed and treated in the two groupsafter the study period of three months. All samples either obtained at home or at the physician's office, will be analyzed by BDProbeTec ET Chlamydia Amplified DNA assay. This is a well documented Nucleid Acid amplification method. Samples will be analysed according to manufactures instructions. Data on number of tested and diagnosed in the two groups will be collected from Stvanger University Hospital. Data on number of treated will be collected from the Norwegain Prescription Database by merging the study dataset with their datafiles. This way we will recive information on who has received treatment for C.rachomatis within one month after after a positive C.trachomatis test.

In Part B a case-cohort from the intervention group (Part A) consisting of a random selection of respondents and non-respondents will be used to determine the feasibility of home sampling as a screening strategy by measuring the risk (OR) related to different factors that determined response. Data are collected through selfadminitered questionnaires.

Part C is a cross sectional study consisting of all respondents in the intervention group. In this part we will measure Prevalence Ratio(PR) of urogential C.trachomatis infections associated with different factors by comparing C.trachomatis positive and C.trachomatis negative in the intervention group.

Part D is an economic study which will be addressed in a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* All persons in the population register in Rogaland County from 18-25 years of age (born between 1/1-1980 - 31/12 -1987) registered 01.11.05. Per 11.11.2005 the size of this population was 41 793. The age cut off is decided because this is the age group with the highest incidence of Chlamydia infections.

Exclusion Criteria:

* All persons in the population register in Rogaland born between 1/1-1980 - 31/12 -1987 registered as:

  * living abroad (including Svalbard) - 6 persons
  * without (permanent) address - 49 persons
  * with client address- 6 persons with secret adress - 16 persons
  * military - 1 person

In total 78 persons were excluded

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41719
Dates: Start 2006-02; Study Completion 2006-09

PRIMARY OUTCOMES:
Yield ratio tested for uro-genital C.trachomatis infection
Yield ratio diagnosed for uro-genital C.trachomatis infection
Yield ratio treated for uro-genital C.trachomatis infection

CONTACTS AND LOCATIONS:
Overall Officials: Preben Aavitsland, MD, Study Director — NIPH
Locations (1):
- Norwegain Institute of Public Health, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Schachter J. Chlamydial infections. West J Med. 1990 Nov;153(5):523-34. No abstract available. PMID 2260289
- [Background] Strand RH, Skjeldestad FE, Ovreness T, Nordbo SA. [Chlamydia trachomatis--pattern of testing and prevalence among young women]. Tidsskr Nor Laegeforen. 2004 Jun 17;124(12):1636-7. Norwegian. PMID 15229709
- [Background] Bakken IJ, Skjeldestad FE, Nordbo SA. [Chlamydia trachomatis infection in women seeking termination of pregnancy 1985-2000]. Tidsskr Nor Laegeforen. 2004 Jun 17;124(12):1638-40. Norwegian. PMID 15229710
- [Background] Andersen B, Olesen F, Moller JK, Ostergaard L. Population-based strategies for outreach screening of urogenital Chlamydia trachomatis infections: a randomized, controlled trial. J Infect Dis. 2002 Jan 15;185(2):252-8. doi: 10.1086/338268. Epub 2002 Jan 3. PMID 11807700
- [Background] van Bergen J, Gotz HM, Richardus JH, Hoebe CJ, Broer J, Coenen AJ; PILOT CT study group. Prevalence of urogenital Chlamydia trachomatis increases significantly with level of urbanisation and suggests targeted screening approaches: results from the first national population based study in the Netherlands. Sex Transm Infect. 2005 Feb;81(1):17-23. doi: 10.1136/sti.2004.010173. PMID 15681716
- [Background] Van Der Pol B, Ferrero DV, Buck-Barrington L, Hook E 3rd, Lenderman C, Quinn T, Gaydos CA, Lovchik J, Schachter J, Moncada J, Hall G, Tuohy MJ, Jones RB. Multicenter evaluation of the BDProbeTec ET System for detection of Chlamydia trachomatis and Neisseria gonorrhoeae in urine specimens, female endocervical swabs, and male urethral swabs. J Clin Microbiol. 2001 Mar;39(3):1008-16. doi: 10.1128/JCM.39.3.1008-1016.2001. PMID 11230419
- [Derived] Klovstad H, Natas O, Tverdal A, Aavitsland P. Systematic screening with information and home sampling for genital Chlamydia trachomatis infections in young men and women in Norway: a randomized controlled trial. BMC Infect Dis. 2013 Jan 23;13:30. doi: 10.1186/1471-2334-13-30. PMID 23343391